CLINICAL TRIAL: NCT01895088
Title: A Continuation Study To Monitor The Long Term Safety Of The AcuFocus ™ ACI 7000PDT Patients Completing Protocols ACU-P08-020/020A
Brief Title: A Continuation Study To Monitor The Long Term Safety Of Patients Completing Protocols ACU-P08-020/020A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACU-P12-020C
Record Dates: First submitted 2013-05-03; First posted 2013-07-10 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Presbyopia
Keywords: presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients prev. impl. with ACI 7000 PDT (Experimental): AcuFocus Corneal Inlay ACI 7000 PDT
  Interventions: Device: AcuFocus Corneal Inlay ACI 7000 PDT

INTERVENTIONS:
Device: AcuFocus Corneal Inlay ACI 7000 PDT — Inlay implanted in cornea for improvement of near vision
  Other Names: AcuFocus KAMRA inlay

SUMMARY:
This is a 2 year follow up study to monitor the long term safety of the ACI 7000PDT in subjects who are still implanted with the ACI and have successfully completed the ACU-P08-020/020A studies.

DETAILED DESCRIPTION:
This is a two year follow up study designed to monitor and obtain long-term safety data of the ACI 7000PDT in subjects who participated and successfully completed the ACU-P08-020/020A studies. Subjects must be able to provide voluntary informed consent, and must sign and be given a copy of the written Informed Consent form prior to participating. This continuation study follows subjects still implanted with the ACI and includes two visits, at 12-month intervals, after subjects have been exited (at Month 36) from the ACU-P08-020/020A studies. The first visit is at Month 48 following implantation followed by a final Month 60 visit. The study parameters being measured at these two visits include:

* Specular microscopy
* Slit lamp and fundus examination (ocular health)
* Corrected and uncorrected visual acuity
* Manifest mid-point refraction
* Corneal topography
* Dry eye assessment
* Mesopic and Photopic contrast sensitivity
* Adverse events and complications

All sites participating in the ACU-P08-020/020A studies were invited to participate in the continuation study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed participation in the ACU-P08-020/020A clinical trial.
* Patients must be able to provide voluntary informed consent, and must sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

* Patients who did not complete ACU-P08-020/020A.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Durrie, M.D., Principal Investigator — Durrie Vision; Chad Betts, M.D., R.Ph, Principal Investigator — MacDonald Eye Associates; Vance Thompson, M.D., Principal Investigator — Vance Thompson Vision; Jay Pepose, M.D., Principal Investigator — Pepose Vision Institute; Kevin Waltz, M.D., Principal Investigator — Eye Surgeons of Indiana; John Vukich, M.D., Principal Investigator — Davis Duehr Dean; Peter Hersh, M.D., Principal Investigator — Cornea and Laser Eye Institute; Thomas Tooma, M.D., Principal Investigator — NVision; Colman Kraff, M.D., Principal Investigator — Kraff Eye Institute; Robert Maloney, M.D., Principal Investigator — Maloney Vision Institute; Scott MacRae, M.D., Principal Investigator — University of Rochester Eye Institute - Strong Vision; Gary Foster, M.D., Principal Investigator — Eye Center of Northern Colorado; Phillip Hoopes, Sr., M.D., Principal Investigator — Hoopes Vision
Locations (13):
- United States (13):
  - McDonald Eye Associates, Fayetteville, Arkansas
  - Maloney Vision, Los Angeles, California
  - NVision, Newport Beach, California
  - Eye Center NOCO, Fort Collins, Colorado
  - Kraff Eye Institute, Chicago, Illinois
  - Eye Surgeons of Indiana, Indianapolis, Indiana
  - Durrie Vision, Overland Park, Kansas
  - Pepose Vision Institute, Chesterfield, Missouri
  - The Cornea & Laser Eye Institute, P.A, Teaneck, New Jersey
  - University of Rochester Eye Institute - Strong Vision, Rochester, New York
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Hoopes Vision, Sandy City, Utah
  - Davis Duehr Dean, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://www.acufocus.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Prev. Implanted With ACI7000PDT: Prev. implanted in ACU-P08-020/020A study
  AcuFocus Corneal Inlay ACI 7000 PDT: corneal inlay
Period: Overall Study
Arm/Group | Patients Prev. Implanted With ACI7000PDT
Started | 271 (1 subject consented for monitoring after device removal (not included in cohort), per FDA request.)
Completed | 253
Not Completed | 18

BASELINE CHARACTERISTICS:
Groups:
- Age, Categorical: Measure Type: Count of Participants
Arm/Group | Age, Categorical
Number analyzed (Participants) | 271
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 271
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 125
Region of Enrollment [Number; unit: participants]
  United States | 271

OUTCOME MEASURES:

1. Primary Outcome: Change (Increase) in Uncorrected Near Visual Acuity
Description: The change in the number of lines of threshold visual acuity achieved postoperatively.
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: lines of visual acuity improvement
Groups:
- Patients Prev. Implanted With ACI7000PDT: Prev. implanted in ACU-P08-020/020A study
  AcuFocus Corneal Inlay ACI 7000 PDT: Inlay implanted in cornea for improvement of near vision
Arm/Group | Patients Prev. Implanted With ACI7000PDT
Number analyzed (Participants) | 271
lines of visual acuity improvement | 3.1 (1.7)

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | Patients Prev. Implanted With ACI7000PDT
Serious Adverse Events (participants affected / at risk) | 10/271
Other Adverse Events (participants affected / at risk) | 23/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Prev. Implanted With ACI7000PDT (N=271)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) — Pontine Hemorrage, Hypertensive Emergency
Carcinoma (General disorders) | 1 (1) — Mucoepidermoid carcinoma of left mandibular gland
Motorcycle Accident (Musculoskeletal and connective tissue disorders) | 1 (1) — Broken collar bone and six broken ribs
Breast Cancer (Reproductive system and breast disorders) | 1 (1)
Joint Replacement Surgery (Surgical and medical procedures) | 3 (3) — Two knee, one hip
Benign Brain Tumor (Surgical and medical procedures) | 1 (1) — Parathyroid gland
Cyst Removal (Surgical and medical procedures) | 1 (1) — Synovial cyst
Appendicitis (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Prev. Implanted With ACI7000PDT (N=271)
Blepharitis (Eye disorders) | 1 (1) — Meibomian gland dysfunction
Secondary Surgical Intervention (Eye disorders) | 4 (4) — Treatment of hyperopic shift - inlay in place (3) Inlay removal
Superficial Punctate Keratitis (Eye disorders) | 1 (1)
Conjunctival cyst (Eye disorders) | 1 (1) — OS
Retinal pigment epithelium granularity (Eye disorders) | 1 (1) — Retinal changes
Corneal abrasion (Eye disorders) | 1 (1) — OS poked by tree branch - resolved in four days
Vision (Eye disorders) | 14 (14) — Decrease in BCDVA two lines at Month 3 or later

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No